CLINICAL TRIAL: NCT06674642
Title: Traditional Indigenous Foods Diet and Health Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA Grand Forks Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: GFHNRC157
Record Dates: First submitted 2024-11-02; First posted 2024-11-05 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Sedentary Behavior; Physical Activity
Keywords: Traditional Indigenous foods diet; American Indians
MeSH Terms: conditions — Sedentary Behavior; Motor Activity

STUDY DESIGN:
Intervention Model Description: The study will employ a single-subject experiment (personalized trial) approach with an ABAB design. The participants will act as their own controls. During Phase A participants will consume their usual (control) diet. During Phase B they will consume a Traditional Indigenous Foods diet provided by the GFHNRC. Randomization in single-subject designs takes the form of random assignment of treatment start times and phase lengths for each participant. Statistical analysis will consist of a mixed model that will be fit with a fixed effect of phase (A1, B1, A2, B2) and random intercept for subject for the for each item being examined.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Traditional Indigenous Foods diet (Experimental): Participants will consume a diet comprised of traditional indigenous foods.
  Interventions: Other: Traditional Indigenous Foods diet

INTERVENTIONS:
Other: Traditional Indigenous Foods diet — A diet composed of traditional indigenous foods will be given to participants.

SUMMARY:
The purpose of this research is to determine whether eating a diet made up of Traditional Indigenous Foods from the Northern Great Plains area will spontaneously result in an increase in physical activity by American Indians, and whether the diet improves metabolic measures of health, mood and self-regulation of healthy eating and engaging in physical activity.

DETAILED DESCRIPTION:
The primary aim of the current study is to determine whether consuming a healthier more Traditional Indigenous Foods diet produces non-targeted simultaneous changes in physical activity of American Indians. Coaction or dual behavior change refers to a spontaneous change in a nontargeted behavior when producing a change in a targeted behavior. A benefit of coactivation is that two healthy behaviors change when targeting just one. Physical activity was chosen as a primary non-targeted behavior because American Indians and Alaska Natives are 34% more likely to report physical inactivity than non-Hispanic Whites. Physical inactivity and sedentary behavior have negative health consequences. Chronic health conditions such as obesity, cardiovascular disease, Type 2 diabetes, and mental health disorders are more prevalent in people who are physically inactive and/or engage in greater sedentary behavior. A unique aspect of the proposed research is that it will develop a traditional indigenous foods diet based on historical research of several tribes (Mandan, Hidatsa, and Arikara (MHA) Nation, Lakota Sioux, Western and Eastern Dakota Sioux, Ojibwa, and Chippewa tribes) that lived in the Northern Great Plains. The nutrient content of the diet will be based on the 2020 Dietary Guidelines for Americans (DGA) Healthy U.S.-Style Dietary Pattern. However, because bovine dairy is not native to the U.S., alternative foods will be used to ensure adequate intake of the nutrients commonly provided by the dairy food groups. Calcium concentration of participants will be carefully monitored. This study will use a personalized trial approach that focuses on understanding individual responses of American Indians living with a heritage from the Northern Great Plains to a Traditional Indigenous Foods diet on behavioral, psychological, and clinical biochemistry outcomes.

ELIGIBILITY:
Inclusion Criteria:

* American Indian
* Body mass index (BMI) of 18.5-42.0 kg/m2

Exclusion Criteria:

* Health condition that impairs mobility or ability to safely be physically active
* Fasting Blood glucose ≥ 126 mg/dl
* Currently taking anti-inflammatory medications
* Pregnant, breast feeding or lactating
* Currently on a regulated diet
* Currently exercising for 60 minutes or longer greater than 2 times per week
* Allergic to any of the study foods shown in the menu and list of ingredients
* Strong aversion to any of the study foods
* Taking one of the following medications: blood thinning drugs, insulin, biologics, chemotherapy or on immune suppressant medications, and those who have started a new hyperglycemic, hypercholesterolemia, anti-depressant, anti-anxiety, or anti-psychotic medication(s) in the last two months.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2024-09-12 (Actual); Primary Completion 2025-04-07 (Actual); Study Completion 2025-04-07 (Actual)

PRIMARY OUTCOMES:
Change in physical activity as measured by Accelerometer | Day 0, Day 7
  Activity will be measured by an accelerometer for seven days in each phase

CONTACTS AND LOCATIONS:
Overall Officials: Julie Hess, PhD, Principal Investigator — USDA Grand Forks Human Nutrition Research Center
Locations (1):
- USDA Grand Forks Human Nutrition Research Center, Grand Forks, North Dakota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Grand Forks Human Nutrition Research Center Current Nutrition Studies — https://www.ars.usda.gov/plains-area/gfnd/gfhnrc/docs/nutrition-studies/nutrition-studies/

DOCUMENTS (1):
  • Informed Consent Form (2024-10-10): https://cdn.clinicaltrials.gov/large-docs/42/NCT06674642/ICF_000.pdf